CLINICAL TRIAL: NCT02875990
Title: Characterization of Immunosuppressive Signing of Cervical Cancer
Acronym: Xac03
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2014-03; 2015-A00699-40 (Registry Identifier: IDRCB)
Record Dates: First submitted 2016-08-12; First posted 2016-08-23 (Estimated); Last update posted 2016-08-23 (Estimated); Status verified 2016-08

CONDITIONS: Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- patients with invasive cervical cancer (Experimental): Blood sample
  Interventions: Biological: Blood sample

INTERVENTIONS:
Biological: Blood sample

SUMMARY:
Infection with Human Papillomavirus high-risk Human (HR-HPV) is the main factor of risk of cancer of the cervix. Recent studies show that cancers linked to infection with HR-HPV are associated with immunosuppression and lack of T cell response Such mechanisms would promote progression to cancer and progression of it . Various factors such as an increase of regulatory T cells, the presence of myeloid cells and suppressor of defects in the signaling pathway Toll Like Receptor (TLR) may have a key role in these immunosuppression mechanisms. At this stage of knowledge, a better characterization of local and systemic immunosuppressive signing of cervical cancer is needed. The results should have a significant medical impact for the identification of new prognostic markers and new therapeutic targets for the treatment of patients with cervical cancer.

The aim of this research project is to define the signing of immunosuppressive cancer cervix and analyze the different mechanisms involved in this immunosuppression.

ELIGIBILITY:
Inclusion Criteria:

* The women presenting for initial therapeutic management of cervical cancer
* Elderly patients over 18 years
* Patients beneficiary of a social security scheme
* Pregnant women can not participate in this study
* Women known to be HIV positive will not participate in this study

Exclusion Criteria:

* Patients with a recurrence of a treaty cervical cancer
* Patients with a history of pelvic radiotherapy
* Patients unable to receive informed about the progress and objectives of the study
* Patients not receiving a social security scheme
* Patients who have not signed informed consent
* Immunocompromised patients and pregnant women

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2016-09; Primary Completion 2024-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Lack of tumor emboli histological analysis | 60 months
  Patients with good prognosis of cervical cancer

CONTACTS AND LOCATIONS:
Locations (1):
- Assistance Publique Hôpitaux de Marseille, Marseille, France

IPD SHARING:
Plan to Share IPD: No